CLINICAL TRIAL: NCT00001455
Title: Iron Overload in African Americans
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950142; 95-CH-0142
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-06

CONDITIONS: Hemochromatosis; Iron Overload
Keywords: Genetics; Hemochromatosis; Iron Metabolism; Iron Storage Disorder; Pedigree; Iron Overload
MeSH Terms: conditions — Hemochromatosis; Iron Overload

SUMMARY:
Iron overload (hemochromatosis) is a condition which causes the intestines to take too much iron into the body from food or pills. The extra iron can build up in the liver, heart, joints, pancreas, sex organs, and other organs. Patients with iron overload can feel well initially, but the iron will eventually damage organs and may lead to an early death. The condition is believed to be passed down from generation to generation. Many studies have been conducted on the condition as it affects Caucasian Americans, few have addressed the condition in African Americans.

Researchers believe it is important to find out as much as possible about the iron overload in African Americans. The goal of this study is to determine the pattern of inheritance of primary iron overload in African American families and to identify the genetic defect causing the condition.

The study will use various tests from simple blood testing (transferritin saturation and serum ferritin levels) to complex genetic tests (segregation analysis and polymerase chain reaction [PCR]). The tests will help researchers deterimine iron levels in the blood, presence of antigens that may help trace inheritance, and detect changes in genes that are known to cause iron overload in Caucasians.

The study may not directly benefit the patients participating in it. However, this study may lead to improved methods to diagnose iron overload in the African American population as a whole.

DETAILED DESCRIPTION:
The purpose of this project is to determine the pattern of inheritance of primary iron overload in African American families and to identify the genetic defect. The iron status of index subjects and family members will be determined by measuring transferrin saturation and serum ferritin, and the genetic pattern will be studied with segregation analysis. The chromosomal localization of the iron-loading locus will be pursued by determining HLA haplotypes, by testing for HFE gene mutations, by sequencing portions of genes for molecules involved in iron metabolism, by analyzing polymorphisms in these genes by PCR, by employing molecular methods to screen the genome, and by testing for linkage to iron phenotype with lod scores. Loci for proteins important in iron metabolism will be examined as candidate genes.

ELIGIBILITY:
Index subjects as well as male and female first and second degree family members, greater than 5 years of age, of index subjects with iron overload.

In some cases, more distant family members will also be studied.

No patients less than or equal to 5 years old.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500
Dates: Start 1995-06; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bassett ML, Halliday JW, Powell LW. Value of hepatic iron measurements in early hemochromatosis and determination of the critical iron level associated with fibrosis. Hepatology. 1986 Jan-Feb;6(1):24-9. doi: 10.1002/hep.1840060106. PMID 3943787
- [Background] Beutler E. The significance of the 187G (H63D) mutation in hemochromatosis. Am J Hum Genet. 1997 Sep;61(3):762-4. No abstract available. PMID 9326341
- [Background] Brink B, Disler P, Lynch S, Jacobs P, Charlton R, Bothwell T. Patterns of iron storage in dietary iron overload and idiopathic hemochromatosis. J Lab Clin Med. 1976 Nov;88(5):725-31. PMID 978039